CLINICAL TRIAL: NCT04531631
Title: Effects of Dorzagliatin on 1st Phase Insulin and Beta-cell Glucose Sensitivity in Individuals With Recent-onset Type 2 Diabetes and Monogenic Diabetes
Brief Title: Effects of Dorzagliatin on 1st Phase Insulin and Beta-cell Glucose Sensitivity in T2D and Monogenic Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CRE-2020.196
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): receive a single oral dose of dorzagliatin 75mg tablet on visit 2 and receive one placebo tablet on visit 3
  Interventions: Drug: Dorzagliatin; Drug: placebo
- Group 2 (Other): receive a single oral dose of one placebo tablet on visit 2 and receive dorzagliatin 75mg tablet on visit 3
  Interventions: Drug: Dorzagliatin; Drug: placebo

INTERVENTIONS:
Drug: Dorzagliatin — tablet
Drug: placebo — placebo

SUMMARY:
Diabetes is a disorder of energy energy metabolism. Glucose is the main energy substrate for generation of ATP to maintain cellular metabolism, structure and function. Glucokinase (GK) serves as a glucose sensor for the initiation of the energy generation.for energy metabolism. Dorzagliatin is a novel, first-in-class, dual-acting allosteric GK activator (GKA). It increases the affinity of GK for glucose by directly binding a pocket distal to its active site, thus lowering the set point for glucose-stimulated insulin secretion in the beta-cell.

Dorzagliatin is a new drug which acts as GK sensor activator (GKA). It can restore the sensitivity of the pancreas cells to glucose and improve glucose control. The drug has been trialled in healthy volunteers and in individuals with type 2 diabetes.

The aim of this study is to understand the way in which dorzagliatin works to improve blood sugar control in people with diabetes. The study will look at how dorzagliatin affects insulin secretion and the sensitivity of the pancreas to changes in blood sugar levels. We will examine whether dorzagliatin can restore the function of this GK sensor in patients with known mutations. In a cross-over study, we will evaluate the effects of dorzagliatin, a specific GKA versus placebo in terms of insulin secretion and beta-cell glucose sensitivity in patients with newly-diagnosed T2D and patients who are known heterozygous carriers of GK mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged ≥ 18 years but < 65years
2. Male or female
3. Body mass index of over 18 kg/m2 and < 30 kg/m2 Additional Inclusion criteria for recent-onset T2D group

   * Diagnosis of T2D for at least 3 months and less than 2 years
   * On diet control only
   * HbA1c>6.5 % and <8% Additional Inclusion criteria for GK MODY-2 group
   * Abnormal fasting plasma glucose >5.6 mmol/l and known heterozygous carrier of pathogenic GK mutation

Exclusion Criteria:

1. Subjects who do not agree to participate in this study.
2. Country of birth is unknown
3. Body weight less than 45kg
4. Acute phase of cerebrovascular and cardiovascular diseases (within 6 months of recruitment).
5. Subjects with severe renal dysfunction as defined by eGFR <30 ml/min/1.73m2 or patients receiving renal dialysis (such as haemodialysis or continuous ambulatory peritoneal dialysis).
6. Severe hepatic dysfunction as defined by AST and/or ALT > 3 times upper limit of normal
7. Severe cardiovascular disease, history of stroke, heart failure (NYHA III or IV) or history of myocardial infarction within last 12 months
8. History of drug abuse or excessive alcohol intake based on investigator judgment
9. Severe hypoglycaemia resulting in seizure/unconsciousness/coma/hospitalization in the last 3 months before screening
10. Diagnosis with Type 1 Diabetes Mellitus (T1DM) or any previous episodes of diabetic ketoacidosis.
11. Dehydration, diarrhoea or vomiting at the time of recruitment
12. Subjects with severe infection, in perioperative period or with serious injury at the time of recruitment
13. Subjects with anaemia (Haemoglobin <9.0mg/dL)
14. Pregnant or lactating or intending to become pregnant within 30 days after last dose of study drug.
15. Participation in a clinical trial within 30 days before enrolment
16. Donation or loss of blood (excluding the volume of blood that will be drawn during screening procedures) as follows: >=300 mL of blood within 30 days prior to study drug administration.
17. Subjects judged unsuitable for the study based on investigator judgment
18. Use of metformin, sulfonylureas, dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 [GLP-1] agonists, sodium glucose transporter 2 inhibitors, insulin, thiazolidinediones, acarbose in the 3 months prior to study enrolment will not be permitted.
19. Use of strong or moderate CYP3A4 inhibitors or inducers and cannot be discontinued
20. Unwilling or unable to follow protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
first phase insulin response to glucose | 10 mins
  measure insulin between 0 to 10 minutes

SECONDARY OUTCOMES:
First phase C-peptide responses to glucose | 10 mins
  measure C peptide between 0 to 10 minutes
Maximum concentration (Cmax) 1st phase insulin between 0 to 10 minutes | 10 mins
  measure insulin between 0 to 10 minutes
Time to maximum (Tmax) of acute phase insulin response between 0 to 10 minutes | 10 mins
  measure insulin between 0 to 10 minutes
Second phase insulin response | 40 mins
  measure insulin at last 40 mins of hyperglycemic clamp
Beta cell glucose sensitivity | 40 mins
  insulin secretion in last 40 minutes of hyperglycemic clamp
Insulin sensitivity index | 40 mins
  glucose infusion rate in last 40 minutes of hyperglycemic clamp
Area under curve of glucagon levels | 120 mins
  measure glucagon from 0-120 mins
Area under curve of GLP-1 levels | 120 mins
  measure GLP-1 from 0-120 mins

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No